CLINICAL TRIAL: NCT03035448
Title: A Randomized Controlled Trial of Communication Strategies to Introduce Psychology Services in the Palliative Care Setting
Brief Title: Communication Strategies to Introduce Psychology Services
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2016-0679; NCI-2018-01285 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2017-01-26; First posted 2017-01-30 (Estimated); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Malignant Neoplasms of Independent (Primary) Multiple Sites
Keywords: Malignant neoplasms of independent (primary) multiple sites; Advanced cancer; Recurrent cancer; Metastatic disease; Palliative care; Videos; Questionnaires; Surveys
MeSH Terms: conditions — Recurrence; Neoplasm Metastasis | interventions — Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video 1: Counselor Alone (Experimental): Participants complete 3 assessment questionnaires during an already-scheduled office visit.
  Participant watches 2 videos showing actors playing a doctor, counselor, and patient, discussing psychology service options.
  Participant completes 3 questionnaires after watching the second video about whether they think 1 of the videos was better than the other, and about their attitude toward psychology services.
  Interventions: Behavioral: Questionnaires; Other: Video Presentation
- Video 2: Doctor + Counselor (Experimental): Participants complete 3 assessment questionnaires during an already-scheduled office visit.
  Participant watches 2 videos showing actors playing a doctor, counselor, and patient, discussing psychology service options.
  Participant completes 3 questionnaires after watching the second video about whether they think 1 of the videos was better than the other, and about their attitude toward psychology services.
  Interventions: Behavioral: Questionnaires; Other: Video Presentation

INTERVENTIONS:
Behavioral: Questionnaires — Participants complete 3 assessment questionnaires during an already-scheduled office visit. These questionnaires should take about 9 minutes to complete.
  Participant completes 3 questionnaires after watching the second video about whether they think 1 of the videos was better than the other, and about their attitude toward psychology services. These questionnaires should take about 4 minutes to complete.
  Other Names: Surveys
Other: Video Presentation — Participant watches 2 videos showing actors playing a doctor, counselor, and patient, discussing psychology service options.

SUMMARY:
The goal of this research study is to learn about advanced cancer patients' preferences about how psychology services are introduced.

This is an investigational study.

Up to 110 participants will be enrolled in this study. All will take part at MD Anderson.

DETAILED DESCRIPTION:
If you agree to take part in this study, during an already-scheduled office visit, you will complete 3 questionnaires about your symptoms, your emotional health, and if you have ever participated in psychiatric or psychology services. These questionnaires should take about 9 minutes to complete.

All participants will watch 2 short videos. The videos show actors playing a doctor, counselor, and patient, discussing psychology service options. Each video is about 1 minute and 30 seconds long and will discuss the same material, but the content of each video will be different. The order in which they are presented will be randomly assigned (as in the flip of a coin). You will have an equal chance of seeing either video first.

After you watch the second video, you will complete 3 questionnaires about whether you think 1 of the videos was better than the other, and about your attitude toward psychology services. These questionnaires should take about 4 minutes to complete.

Length of Study:

It should take about 16 minutes to watch both videos and to complete all questionnaires. Your participation on this study will be over after you have completed the last questionnaire.

Other Information:

We will ask your caregiver(s) to leave the room while the videos are played. In case they decide to stay, we will ask them to keep silent.

ELIGIBILITY:
Inclusion Criteria:

1. Age >/= 18 years-old
2. Can speak, read, and understand English
3. Diagnosis of locally advanced, recurrent, or metastatic disease
4. Patients treated as outpatients by the supportive and palliative care team
5. Normal cognitive status as determined by the interviewer based on the ability to understand the nature of the study and consent process

Exclusion Criteria:

1. Previous psychological counseling received in supportive care department
2. Patients with severe symptom distress as assessed by nursing staff

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2017-02-13 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2023-10-10 (Actual)

PRIMARY OUTCOMES:
Participant's Video Preference of Strategies in Introducing Psychology Services in a Palliative Care Setting | Day 1
  Participants asked the preference to the introduction of counselor. The possible answers are The First Video, The Second Video, Neither, or No Difference. The actual content of the answers will be decoded by the study team at the end of the study to "Counselor Alone" or "MD + Counselor" depending on each patient's assigned arm.

CONTACTS AND LOCATIONS:
Overall Officials: Sujin Ann-Yi, PHD, MA, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org